CLINICAL TRIAL: NCT05312138
Title: The Effect of Different Neuromodulation Techniques in the Treatment of Multiple Sclerosis Patients With Neurogenic Bladder Dysfunction
Brief Title: Multiple Sclerosis and Overactive Bladder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, pnaratak, assistant professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: patak
Record Dates: First submitted 2021-12-26; First posted 2022-04-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Neurogenic Bladder Dysfunction
Keywords: Multiple Sclerosis; Overactive Bladder; Neurogenic Bladder; Electrical stimulation
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive; Urinary Bladder, Neurogenic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Posterior Tibial Nerve Stimulation Group (Experimental): The treatment will be carried out by the physiotherapist using the TenStem Eco Basic device.
  Interventions: Device: Transcutaneous Posterior Tibial Nerve Stimulation
- Repetitive Transcranial Magnetic Stimulation Group (Active Comparator): The treatment will be applied with a Power Mag device.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The treatment will be internally cooled 70 mm double coil and 110 mm round coil, accompanied by a physiotherapist and neurologist. The coil will be placed on the precentral gyrus. Practices will be held, with each session lasting 20 minutes. Cortical excitability will be provided by high frequency (HF) stimulation (5-Hz).
  Arms: Repetitive Transcranial Magnetic Stimulation Group
Device: Transcutaneous Posterior Tibial Nerve Stimulation — The treatment parameters will be applied with a pulse current time of 200 μsec, a fixed frequency of 10 Hz, a treatment time of 20 minutes, and a current intensity that the patient can tolerate, which will not cause flexion in the big toe or fan movement in the other fingers. Self-adhesive surface electrodes will be used for stimulation. During the treatment, the patient will lie on his back. The negative electrode will be placed 2 cm posterior to the medial malleolus and the positive electrode will be placed 10 cm proximal.
  Arms: Transcutaneous Posterior Tibial Nerve Stimulation Group

SUMMARY:
Urinary symptoms are frequently seen in patients with Multiple Sclerosis (MS). Early evaluation of the patients in terms of the urinary system, planning the appropriate treatment and following up at regular intervals are extremely important in terms of preventing urinary system complications. Neuromodulation applications are used reliably in the urological treatment of MS patients. The aim of this study was to compare the efficacy of different neuromodulation techniques, transcutaneous posterior tibial nerve stimulation and repetitive transcranial magnetic stimulation, in patients with MS reporting lower urinary tract symptoms.

DETAILED DESCRIPTION:
Bladder dysfunction is one of the most disturbing symptoms of MS. The frequency of bladder dysfunction in patients with MS is reported to be %52-97. Urinary symptoms are among the initial symptoms in %10-15 of patients, while it is the only initial symptom in up to %2 of patients. Patients is seen with irritative symptoms (such as frequent urination, urgency, urinary incontinence, nocturia), obstructive symptoms (such as difficulty in initiating urination, inability to urinate, feeling of incomplete emptying, weak urine flow) or mixed type symptoms.In line with these symptoms, early evaluation of MS patients in terms of urinary system, planning of appropriate treatment and regular follow-up are extremely important in terms of preventing urinary system complications. Pharmacotherapy and clean intermittent catheterization are the first step treatments for lower urinary tract symptoms in multiple sclerosis. It has been reported in the literature that electrical nerve stimulation therapy (neuromodulation methods) and behavior change methods (pelvic floor muscle exercise, bladder training, urinary diary keeping) are also used as a second step treatment option due to the side effects of anticholinergic use and lack of motivation and skill in catheterization. It is reported that neuromodulation applications are performed in MS patients and it is a reliable method. Deep brain stimulation, transcranial magnetic stimulation, posterior tibial nerve stimulation, sacral neuromodulation and spinal cord stimulation are generally recommended in the treatment of bladder dysfunction, which is one of the neuromodulation methods. The superiority of these methods to each other is debatable. In line with this information, the aim of the study is to compare the effectiveness of different neuromodulation techniques, transcutaneous posterior tibial nerve stimulation and repetitive transcranial magnetic stimulation, in MS patients reporting lower urinary tract symptoms.

According to the treatment protocols of the patients to be included in the study; will be divided into 2 groups as transcutaneous posterior tibial nerve stimulation group (8 patients) and repetitive transcranial magnetic stimulation group (8 patients). Which method will be applied to which individual will be determined randomly. Treatment sessions will be carried out for 5 consecutive days in 2 consecutive weeks, 1 time per day for a total of 10 sessions. The urological parameters of the patients in all groups will be evaluated before and after the treatment.

Statistical method(s); Statistical analysis of the data obtained from the study will be done in the Statistical Package for the Social Sciences (SPSS) 22.0 package program. The mean standard deviation, median, minimum and maximum values will be used to define the data. Comparison of continuous variables between groups will be done with Mann Whitney U test, comparison of discrete variables will be done with chi-square test. Spearman or Pearson correlation test will be used to evaluate the correlation between variables. In the data analysis, p < 0.05 level will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Woman
* Volunteer to participate in the study
* Neurogenic overactive bladder due to MS
* EDSS <7.0
* Not benefiting from pharmacological treatment

Exclusion Criteria:

* With urinary tract infection
* Diagnosed with diabetes mellitus
* Using diuretic medication
* Using clean intermittent catheterization
* Having a history of different urological diseases
* Those who have conditions that would be contraindicated for electrical stimulation (pacemaker, brain pacemaker, prosthesis)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Urodynamics Test | "10 days" the amount of change after 10 days from the baseline
  While the bladder is being filled, it will be carried out to measure the pressures in the bladder and in the abdomen, to examine the nerves that provide bladder contractions, and to explain the cases of urinary incontinence or inability by examining the bladder contraction pressures and electrical activity during urination.
Extended Disability Status Scale (EDSS) | "10 days" the amount of change after 10 days from the baseline
  It is the most commonly used scale to assess disability in MS. EDSS scoring is based on the neurological examination results of eight functional systems and the patient's ambulation status. Functional systems are listed as pyramidal, cerebellar, brainstem, sensory, bladder and intestinal, visual, cerebral, and others. A score of 0-10 is given.0 denotes normal neurological examination, 10 denotes death due to MS. 1.0-4.5 refers to fully ambulatory, 5.0-9.5 refers to impaired ambulation. From 7.0 onwards there is wheelchair use and increasingly bed dependency.
Overactive Bladder Questionnaire-V8 (OAB-V8) | "10 days" the amount of change after 10 days from the baseline
  The severity of the patients' complaints, none (0); very few (1); a little (2); quite a few (3); many (4); and too many (5) it consists of 8 questions that can be graded. The total score can vary between 0 and 40.
Incontinence Quality of Life -I-QOL | "10 days" the amount of change after 10 days from the baseline
  It consists of a total of 22 questions with three sub-dimensions. Sub-dimensions; limitation of behaviors (1,2,3,4,10,11,13,20 items), psychosocial influence (5,6,7,9,15,16,17,21,22 items) and social isolation (8,12 ,14,18,19 items). All items are evaluated with a five-point Likert type (1= too much, 2= a quite, 3= moderately, 4= a little, 5= not at all) and the Likert types are recalculated to take a value between 0-100 points in order to better understand the total score calculated. Higher scores indicate better quality of life.
Voiding Diary | "10 days" the amount of change after 10 days from the baseline
  It is recommended to present the information given by the patients in an objective way. Although not entirely diagnostic, diary data can reveal normal and abnormal conditions. The 3-day voiding diary is a viable, reliable and valid tool in the evaluation of patients with lower urinary tract symptoms.
Incontinence Severity Index (ISI) | "10 days" the amount of change after 10 days from the baseline
  It consists of 2 questions, and the total score is obtained by multiplying the frequency of urinary incontinence and the amount of urine leaked, and the score range varies between 1-12. According to their score, 1-2 points are light; 3-6 points average; 8-9 points indicate severe and 12 points very severe urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Atak Çakır, Principal Investigator
Locations (1):
- Istanbul Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No Plan Description

REFERENCES:
- [Background] Nardone R, Versace V, Sebastianelli L, Brigo F, Golaszewski S, Christova M, Saltuari L, Trinka E. Transcranial magnetic stimulation and bladder function: A systematic review. Clin Neurophysiol. 2019 Nov;130(11):2032-2037. doi: 10.1016/j.clinph.2019.08.020. Epub 2019 Sep 3. PMID 31541980
- [Background] de Seze M, Raibaut P, Gallien P, Even-Schneider A, Denys P, Bonniaud V, Game X, Amarenco G. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. Neurourol Urodyn. 2011 Mar;30(3):306-11. doi: 10.1002/nau.20958. Epub 2011 Feb 8. PMID 21305588
- [Background] Abboud H, Hill E, Siddiqui J, Serra A, Walter B. Neuromodulation in multiple sclerosis. Mult Scler. 2017 Nov;23(13):1663-1676. doi: 10.1177/1352458517736150. PMID 29115915
- [Background] Fingerman JS, Finkelstein LH. The overactive bladder in multiple sclerosis. J Am Osteopath Assoc. 2000 Mar;100(3 Suppl):S9-12. PMID 10763312
- [Derived] Atak Cakir P, Guzelburc V, Birday E, Hanoglu L, Mutluay F. Effect of neuromodulation on neurogenic bladder in women with multiple sclerosis: a pilot randomized controlled trial. Neurodegener Dis Manag. 2025 Apr-Jun;15(2-3):57-64. doi: 10.1080/17582024.2025.2488712. Epub 2025 Apr 11. PMID 40211880
- [Derived] Atak Cakir P, Mutluay F, Hanoglu L, Guzelburc V. Effect of transcutaneous posterior tibial nerve stimulation and repetitive transcranial magnetic stimulation on neurogenic overactive bladder symptoms in female patients with multiple sclerosis: The study protocol of a randomized controlled study. Front Neurol. 2022 Oct 28;13:1011502. doi: 10.3389/fneur.2022.1011502. eCollection 2022. PMID 36388236

DOCUMENTS (3):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05312138/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05312138/SAP_001.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT05312138/ICF_002.pdf